CLINICAL TRIAL: NCT01035008
Title: Detection of Neoplastic Pancreatic Cysts Using Probe Based Confocal Laser Endomicroscopy: A Prospective in Vivo Study
Brief Title: Confocal Endomicroscopy of Pancreatic InVivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Mauna Kea Technologies (Industry)
Responsible Party: Michael B. Wallace, MD MPH, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-006345
Record Dates: First submitted 2009-12-04; First posted 2009-12-18 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Pancreatic Cysts
Keywords: pancreatic cysts
MeSH Terms: conditions — Pancreatic Cyst | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Microscopy, Confocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (Experimental): The investigators are testing a new method called confocal laser endomicroscopy to see if it can detect pre-cancerous abnormalities in the lining of the cysts found in your pancreas. This will involve using a very thin fiber-shaped microscope which will be passed through a needle during the EUS procedure.
  Interventions: Procedure: Endoscopic Ultrasound (EUS)

INTERVENTIONS:
Procedure: Endoscopic Ultrasound (EUS) — The investigators will do the standard EUS procedure. If a cyst is seen in the pancreas during EUS, the investigators will administer a special dye called fluorescein through the IV, and then use the new fiber-shaped microscope to take pictures of the lining of the cysts.
  Other Names: Cellvizio Endomicroscopy; Confocal; Endoscopic Ultrasound

SUMMARY:
Confocal laser endomicroscopy (CLE) is a novel and highly promising imaging method for that allows in vivo imaging of the mucosal layer at resolution of approximately 1 micron. Cellular and sub-cellular structures as well as capillaries and single red blood cells can be visualized. CLE is now well established as a highly accurate method for distinguishing neoplasia in the gastrointestinal tract lumen via endoscopy. A major new breakthrough is the development of sub-millimeter CLE probes that can be passed via an image guided needle (nCLE) into solid organs and cysts.

It is hypothesized that nCLE will help distinguish the benign, premalignant and malignant cystic lesions of pancreas by visualizing the cellular lining of the cysts, thereby, avoiding unnecessary surgery in patient with benign cysts and guiding to early and effective surgical removal of high risk neoplastic lesions.

A prototype minimal risk nCLE system has been developed that can be passed via standard endoscopic ultrasound needles into the pancreas but FDA clearance for in vivo use is not expected until late 2010. The investigators propose to evaluate this prototype nCLE system in vivo during endoscopic ultrasound (EUS), as an initial pilot study.

DETAILED DESCRIPTION:
Hypothesis: the confocal laser endomicroscopy imaging of the nCLE can differentiate between non-mucinous, mucinous non- malignant and malignant pancreatic cysts in vivo and has increased sensitivity compared to endoscopic ultrasound-fine needle aspiration (EUS-FNA) tissue sampling. In this pilot study the investigators will primarily evaluate technical feasibility and interobserver agreement.

1. In patients undergoing EUS for suspected pancreatic cysts, the investigators will evaluate the key nCLE image features of non mucinous, mucinous, and malignant pancreatic cystic neoplasms (PCN).
2. The investigators will estimate the initial image quality, feasibility, and interobserver agreement of nCLE
3. The investigators will establish the preliminary accuracy of nCLE to be used for planning a larger comparative trial

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing endoscopic ultrasound for evaluation of pancreatic cysts (including pseudocysts and suspected pancreatic cystic neoplasms) in the gastrointestinal (GI) lab at Mayo Clinic Jacksonville.

Exclusion Criteria:

* Unwilling/unable to consent;
* Solid pancreatic mass on computerized axial tomography/magnetic resonance (CT/MR);
* Allergy to Fluorescein;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Differentiate between non-mucinous, mucinous non-malignant & malignant pancreatic cysts in vivo | One day (completion of the EUS)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Wallace, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States